CLINICAL TRIAL: NCT00201435
Title: Weekly Taxol® Plus Xeloda® Versus Taxotere® Every Three Weeks Plus Xeloda® in the Treatment of Metastatic Breast Cancer A Phase II/III Study
Brief Title: Weekly Taxol Plus Xeloda® vs Taxotere q3wk Plus Xeloda® in the Treatment of Metastatic BC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Norwegian Breast Cancer Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBCG10; REK 378-04-03133; NMA 03-07568
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Breast Neoplasm
Keywords: Breast; Cancer; Paclitaxel; Docetaxel; Qulaity of life
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Paclitaxel weekly in combination with capecitabine
Drug: Docetaxel every 3 week in combination with capecitabine

SUMMARY:
We want to compare Taxol given weekly with Taxotere given every 3 week both in comination with Xeloda. We are going to compare time to treatment failure and quality of life.

DETAILED DESCRIPTION:
Open labeled randomized multicentre phase II/III trial. It is intended to include patients who are not usually included into clinical trials because they are not having disease with measurable lesions. In breast cancer the bulk of patients with metastatic disease is presenting with bone metastases which is difficult to evaluate with respect to response. In this study it is one of the main objectives to include this kind of everyday patients that we see in the clinic.

Because of this we will be using TTF as the primary endpoint. Skeletal events requiring radiotherapy or major changes in pain medications are defined as treatment failures causing stop in treatment even in the absence of radiological findings.

A: weekly Taxol® plus Xeloda® on days 1-14 q 3w B: Taxotere® q 3w plus Xeloda® on days 1-14 q 3w

Patients are randomized equally between the two arms.

Concomitant therapy: Simultaneous use of bisphosphonates is allowed, if this treatment has been initiated at least four weeks before study entry.

ELIGIBILITY:
Inclusion Criteria: Morphologically proven breast carcinoma

Written informed patient consent Measurable and/or evaluable disease Measurable disease is defined as least one lesion that can be accurately measured in at least one dimension as ≥20 mm by conventional techniques, or as ≥10 mm by spiral CT scan) as defined in section 8.

Evaluable metastases. Lytic bone metastases as only site of recurrence are allowed and can be evaluated for response according to the WHO-criteria for reporting on response in bone metastases.

Age 18 years or older ECOG Performance Status 0-2 Life expectancy of at least three months Adequate cardiac functions

Adequate hematological, renal and hepatic functions, defined as:

White blood cell count > 3.9 x 109/L Trombocytes > 100 x 109/L Serum creatinine < 1.25 x ULN* Bilirubin < 1.5 ULN If alkaline phosphatases (ALP) is normal ALAT < 3.5 ULN ASAT < 3.5 ULN If alkaline phosphatases (ALP) is > 2.5 ULN ALAT < 1.5 ULN ASAT < 1.5 ULN

-

Exclusion Criteria: Recurrence-free interval less than one year, if previous adjuvant or neoadjuvant regimen contained a taxane

Neoplasm other than breast carcinoma, except for non-melanoma skin cancer or curatively treated carcinoma in situ of the cervix, diagnosed during the past five years

Pregnancy or lactation

Known brain metastases

Preexisting motor or sensory neuropathy ≥ grade 2 according to NCI CTC 2.0 criteria (severe paresthesia and/or mild weakness, or worse)

Severe hepatic or renal impairment (for capecitabine: calculated creatinine clearance below 30 ml/min; for calculation, see p. 5.1.4) not allowing for adequate use of the proposed regimens

History of known dihydropyrimidine dehydrogenase (DPD) deficiency (severe reaction on previous treatment with fluorouracil)

Active infection or other serious underlying medical condition which would impair the ability of the patient to receive protocol treatment, including prior allergic reactions to drugs containing cremophor, such as teniposide, cyclosporine or vitamin K

Dementia or significantly altered mental status that would prohibit the understanding and giving of informed consent.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2005-03; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure
Quality of life

SECONDARY OUTCOMES:
Response rates
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Erik Wist, MD, PhD, Principal Investigator
Locations (1):
- Ullevål university hospital, Oslo, Norway